CLINICAL TRIAL: NCT04324632
Title: Role of Magnetic Resonance Enterography (MRE) in Assessment of Inflammatory Bowel Diseases.
Brief Title: Magnetic Resonance Enterography in Inflammatory Bowel Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hayam Yahia Hmed Khalil, principal invistigator, Assiut University
Other Study IDs: MRE in IBD
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Inflammatory Bowel Diseases
Keywords: MRE
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assess the accuracy of magnetic resonance-enterography in predicting the extension, location and characteristics of the small bowel segments affected by Crohn's disease& determine the diagnostic performance of standard MR enterography in detecting colonic inflammation and investigate MR enterography's ability to grade inflammatory activity and detect intestinal extra intestinal manifestations

DETAILED DESCRIPTION:
Inflammatory bowel diseases (IBD) are chronic disorders of the gastrointestinal tract with a remitting-relapsing disease pattern. Ulcerative colitis (UC) and Crohn's disease (CD) represent the two main forms of IBD.

In CD inflammation affects various parts of the bowel, separated by unchanged intestinal segments, while in ulcerative colitis enteric involvement is continuous, extending from the rectum throughout the colon. Additionally, in Crohn's disease the inflammatory process spreads through all layers of the intestinal wall, while in UC only the mucosa and sub mucosa are affected.

Imaging findings, endoscopic studies and histological data together with clinical assessment, can be used to help distinguish these two forms, determine prognosis, assess disease activity and to inform treatment decision-making.

A "treat-to-target" strategy with close monitoring of intestinal inflammation is recommended in inflammatory bowel disease (IBD). Ileocolonoscopy (CS) remains the gold-standard for assessing disease activity in IBD but is a relatively invasive procedure and is impossible to repeat in the context of tight monitoring strategies.

MRE is preferred over computed tomography enterography by most radiologists and gastroenterologists because of the potential for differentiating active inflammation from fibrotic strictures, and due to the lack of exposure to ionizing radiation. This is especially true in children, as the onset of IBD in childhood is a known risk factor for high cumulative exposure to ionizing radiation from imaging.

MRE furthermore provides a transmural study of bowel loops (oedema, wall thickening, and enhancement post contrast). These features make MRE ideally suitable to the IBD population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with different age groups and both sex are eligible for our prospective study

  1. Either they had undergone colonoscopy or colonoscopy was planned, and they have been recently diagnosed with IBD.
  2. Suspected to have disease relapse.

Exclusion Criteria:

Participants are not eligible for our prospective study if they:

1. Have evidence of severe or uncontrolled systemic disease that rendered the individual unsuitable for participation.
2. Have contraindications to MRE (e.g. allergy to all suitable contrast agents, cardiac pacemaker, severe claustrophobia, an inability to lie flat).
3. Had a final diagnosis other than IBD.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: subjects of both sexes with different age groups diagnosed to have inflammatory bowel disease
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
comparison of magnetic resonance enterography findings with colonoscopic findings and clinical activity scores of IBD | two years
  To investigate MR enterography's ability to detect to the extension, location and characteristics of intestinal segments affected by IBD and grade inflammatory activity in correlation with endoscopic findings.